CLINICAL TRIAL: NCT05902429
Title: Effects of Oral Cladribine on Remyelination and Inflammation in Multiple Sclerosis Patients
Acronym: CLAREMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Merck S.A., Brazil, an affiliate of Merck KGaA, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS700568_0128
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis; cladribine tablets; remyelination
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Cladribine; Tablets

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, phase IV, single-center, proof-of-concept clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cladribine tablets (Experimental)
  Interventions: Drug: Cladribine 10 mg oral tablet

INTERVENTIONS:
Drug: Cladribine 10 mg oral tablet — Cladribine tablets (Mavenclad®, Merck KGaA, Darmstadt, Germany) will be given according to the label with a cumulative dose of 3.5 mg/kg body weight distributed over 2 years as one treatment course of 1.75 mg/kg per year. Each treatment course will consist of 2 weeks of treatment, one at the beginning of the first month and one at the beginning of the second month of the respective year of treatment. Each treatment week will consist of 4 or 5 days in which the participant will receive 10 mg or 20 mg (1 or 2 tablets, respectively) as a single daily dose, depending on body weight, according to the tables available in label. Upon completion of the two treatment courses, no further courses will be required in years 3 and 4.
  Other Names: Mavenclad

SUMMARY:
Multiple sclerosis (MS) is a chronic, immune-mediated, demyelinating disease of the central nervous system. Typical brain lesions of the disease may be partially repaired by an endogenous remyelination process which is limited and tends to deplete over the course of the disease. Cladribine tablets are an approved treatment that promotes selective lymphocyte depletion, reducing the inflammatory activity of the disease. The present study is based on the hypothesis that improved inflammatory control through cladribine tablets provides a tissue microenvironment more favorable for remyelination of brain lesions in MS. This hypothesis will be evaluated by a single-arm, open-label, phase IV, single-center, proof-of-concept clinical trial in which 10 participants with relapsing-remitting, highly active MS, relatively early in the course of the disease, will receive conventional treatment with cladribine tablets and will be followed-up for 48 months. Neurological, neuropsychological and magnetic resonance imaging (MRI) parameters will be measured. Remyelination will be assessed by a novel MRI technique called the q-Space myelin map. Additionally, the peripheral blood lymphocyte and cytokine profiles will be evaluated in order to understand the immunological aspects that influence the remyelination capacity in patients treated with cladribine tablets. The study will be conducted in accordance with current regulations governing clinical research in Brazil.

ELIGIBILITY:
Inclusion criteria:

Participants who meet all of the following criteria will be included:

* Consent to participate in the study by signing the ICF;
* Age between 18 and 55 years, inclusive;
* Relapsing-remitting multiple sclerosis diagnosed according to 2017 revised McDonald's criteria;
* Highly active disease, defined as 1) occurrence of ≥2 relapses within 12 months prior to study enrolment, regardless of whether or not treatment with another disease-modifying drugs (DMD) was present; or 2) occurrence of ≥1 relapse in the previous 12 months during treatment with another DMD, together with ≥1 gadolinium-enhanced T1 lesion or ≥9 T2/FLAIR lesions on MRI performed during the same period;
* Disease duration (time since first relapse) ≤4 years;
* EDSS score ≤5.0;
* Eligibility for treatment with cladribine tablets, according to the label approved in Brazil;
* For women or men of childbearing potential: agreement to use effective contraceptive method as recommended in cladribine tablets label.

Exclusion criteria:

Participants who meet any of the following criteria will be excluded:

* Contraindications to the use of cladribine tablets (as per the label), including (but not limited to) baseline lymphopenia (<1,000 cells/ mm³), active neoplasm or neoplasm within the last 5 years, active infections (especially tuberculosis, hepatitis B or C and HIV), latent tuberculosis without proper treatment, moderate to severe renal or hepatic impairment, use of immunosuppressants or immunosuppression for another cause;
* Pregnancy or lactation;
* Presence of other medical conditions or current or previous use of another therapy capable of interfering with neurological, neuropsychological, radiological or laboratory evaluation, as per investigator's judgment;
* Contraindications to MRI or gadolinium use;
* Inability to adhere to study procedures, as per investigator's judgment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of remyelinated lesions (as assessed by neuroradiologist) in q-Space myelin map | 36 months after initiation of cladribine tablets treatment

SECONDARY OUTCOMES:
Median "lesion ratio" (i.e., myelin index: lesion signal / normal appearing white matter signal) in q-Space myelin map | 36 months after initiation of cladribine tablets treatment
Mean signal intensity of lesions in q-Space myelin map | 36 months after initiation of cladribine tablets treatment
Correlation between lymphocyte profile and remyelination parameters in q-Space myelin map | Transversally (at months 0, 12, 24, and 36) and longitudinally (over 36 months following initiation of cladribine tablets treatment)
Correlation between cytokine profile and remyelination parameters in q-Space myelin map | Transversally (at months 0, 12, 24, and 36) and longitudinally (over 36 months following initiation of cladribine tablets treatment)
Correlation between remyelination parameters in q-Space myelin map and evolution of clinical scores (annualized relapse rate, EDSS, MSFC and their subtests) | Over 36 months following initiation of cladribine tablets treatment
Correlation between remyelination parameters in q-Space myelin map and evolution of neuropsychological scores (BICAMS and MFIS subtests) | Over 36 months following initiation of cladribine tablets treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Pontifical Catholic University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No